CLINICAL TRIAL: NCT01027273
Title: Preventing Recurrence of All Inner-city Strokes Through Education
Brief Title: Prevent Return of Stroke Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); North General Hospital, New York (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 02-0515 Project 1; 5P60MD000270-08 (NIH)
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Stroke Recurrence; Transient Ischemic Attack
Keywords: Stroke; Ischemic Stroke; Transient Ischemic Attack; Stroke Recurrence Prevention; Cerebrovascular Disorders; Brain Ischemia; Brain Infraction; Brain Diseases; Cerebral Infraction; Self-management; Peer-led; Community Based
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke; Ischemic Stroke; Cerebrovascular Disorders; Brain Ischemia; Brain Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer-Led Stroke Recurrence Prevention Education (Experimental): The intervention group will participate in a 6-session course held over a 6-week period. The Prevent Return of Stroke Workshop, led by trained peer educators, aims to help participants control the risk factors for stroke, thereby preventing recurrence of strokes.
  Interventions: Behavioral: Prevent Return of Stroke
- Usual Care (Delayed Intervention) (Placebo Comparator): The control group will be offered the chance to take part in the 6-week session intervention after 12 months after enrollment into the trial.
  Interventions: Behavioral: Prevent Return of Stroke

INTERVENTIONS:
Behavioral: Prevent Return of Stroke — Prevent Return of Stroke is a community-based, peer-led stroke recurrence prevention program. This is a bilingual (English/Spanish) education program written at a 4th grade reading level, and contains simple, actionable, messages, easily taught by lay leaders, and focuses on enhancing self-efficacy to make lifestyle changes, to help reduce stroke recurrence risk factors. It consists of 6 sessions (1½ hours each) held over 6-weeks. Topics include learning the risk factors for stroke, controlling hypertension, LDL cholesterol, preventing blood clots, medication adherence, and stress management.The intervention arm will participate in the intervention shortly after enrolling in the trial.
  Arms: Peer-Led Stroke Recurrence Prevention Education
Behavioral: Prevent Return of Stroke — The intervention arm will participate in the intervention shortly after enrolling in the trial. The usual care arm will be offered the intervention after 12 months from enrolling in the trial.
  Arms: Usual Care (Delayed Intervention)

SUMMARY:
The purpose of this study is to evaluate if a peer-led stroke recurrence prevention intervention, versus usual care, will help reduce risk factors for recurrent strokes among adults in Harlem.

DETAILED DESCRIPTION:
Twenty nine percent of the 700,000 strokes that occur yearly nationwide are among stroke survivors. Blacks, both nationally and among Harlem residents, have a twofold increase in recurrent strokes. Harlem Latinos have a threefold increase in risk relative to Whites.

Primary risk factors for recurrent stroke include hypertension, hyperlipidemia, and under use of anti-thrombotic agents. Controlling risk factors can be particularly challenging for low-income, minority populations who lack the resources needed to adhere to necessary therapies. In Harlem, 72% of adults studied six months post stroke did not have these three risk factors treated adequately.

We propose to determine if participation in a recurrent stroke prevention educational intervention, versus usual care, can activated stroke survivors to at reduce primary risk factors for recurrent strokes while providing an effective, low-cost, sustainable recurrent stroke prevention program in neighborhoods like Harlem, whose residents bear a disproportionate burden of suffering from strokes. Specifically, we propose:

1. Recruit 600 adults who sustained a stroke or transient ischemic attack (TIA) within the past five years by working with Harlem community leaders, local clinical sites including the Mount Sinai Medical Center and the Institute for Family Health, and the Visiting Nurse Service of New York;
2. To conduct a randomized, controlled trial to determine if participation in a peer-led stroke prevention program activates stroke and TIA survivors to improve their knowledge and self-management strategies and treatments related to stroke prevention; and
3. To rigorously compare the impact of the intervention with usual care (delayed intervention), on increasing the proportion of individuals with strokes and TIAs who are appropriately treated to reduce the risk of recurrent events, specifically through control of hypertension (blood pressure ≤ 140/90mmHg), hyperlipidemia (LDL cholesterol≤100 mg/dl) and use of anti-thrombotic medicines.

ELIGIBILITY:
Inclusion Criteria:

* Had a stroke or TIA diagnosed within 5 years
* 40 years of age or older
* Able to participate in group education classes
* English or Spanish speaking
* Community dwelling

Exclusion Criteria:

* No incidence of stroke or TIA
* Stroke or TIA occurred more than 5 years ago
* less than 40 years of age
* Cognitive or physical impairment that would preclude comprehension of a conversation and communicating as part of a group (i.e., dementia, deafness, inability to speak, aphasia)
* Self-reported terminal illness with life expectancy of less than 1 year
* Plans to relocate from New York City within one year of enrollment
* Pregnant
* Nursing home resident
* Prisoner

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2009-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol R Horowitz, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Goldfinger JZ, Kronish IM, Fei K, Graciani A, Rosenfeld P, Lorig K, Horowitz CR. Peer education for secondary stroke prevention in inner-city minorities: design and methods of the prevent recurrence of all inner-city strokes through education randomized controlled trial. Contemp Clin Trials. 2012 Sep;33(5):1065-73. doi: 10.1016/j.cct.2012.06.003. Epub 2012 Jun 15. PMID 22710563
- [Background] Kronish IM, Edmondson D, Goldfinger JZ, Fei K, Horowitz CR. Posttraumatic stress disorder and adherence to medications in survivors of strokes and transient ischemic attacks. Stroke. 2012 Aug;43(8):2192-7. doi: 10.1161/STROKEAHA.112.655209. Epub 2012 May 22. PMID 22618380
- [Background] Kronish IM, Diefenbach MA, Edmondson DE, Phillips LA, Fei K, Horowitz CR. Key barriers to medication adherence in survivors of strokes and transient ischemic attacks. J Gen Intern Med. 2013 May;28(5):675-82. doi: 10.1007/s11606-012-2308-x. Epub 2013 Jan 4. PMID 23288379
- [Background] Edmondson D, Horowitz CR, Goldfinger JZ, Fei K, Kronish IM. Concerns about medications mediate the association of posttraumatic stress disorder with adherence to medication in stroke survivors. Br J Health Psychol. 2013 Nov;18(4):799-813. doi: 10.1111/bjhp.12022. Epub 2013 Jan 7. PMID 23294320
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Kronish IM, Goldfinger JZ, Negron R, Fei K, Tuhrim S, Arniella G, Horowitz CR. Effect of peer education on stroke prevention: the prevent recurrence of all inner-city strokes through education randomized controlled trial. Stroke. 2014 Nov;45(11):3330-6. doi: 10.1161/STROKEAHA.114.006623. Epub 2014 Sep 23. PMID 25248910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from June 2009 to June 2012 recruited at community based sites as well as clinical sites.
Groups:
- Peer-Led Stroke Recurrence Prevention Education: The intervention group participated in a 6-session course held over a 6-week period. The Prevent Return of Stroke Workshop, led by trained peer educators, aimed to help participants control the risk factors for stroke, thereby preventing recurrence of strokes.
  Prevent Return of Stroke: Prevent Return of Stroke is a community-based, peer-led stroke recurrence prevention program. This is a bilingual (English/Spanish) education program written at a 4th grade reading level, and contains simple, actionable, messages, easily taught by lay leaders, and focuses on enhancing self-efficacy to make lifestyle changes, to help reduce stroke recurrence risk factors. It consists of 6 sessions (1½ hours each) held over 6-weeks. Topics include learning the risk factors for stroke, controlling hypertension, LDL cholesterol, preventing blood clots, medication adherence, and stress management.The intervention arm will participate in the intervention shortly after enrolling in the trial.
- Usual Care (Delayed Intervention): The control group was offered the chance to take part in the 6-week session intervention after 12 months after enrollment into the trial.
  Prevent Return of Stroke: The intervention arm participated in the intervention shortly after enrolling in the trial. The usual care arm was offered the intervention after 12 months from enrolling in the trial.
Period: Overall Study
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Started | 301 | 299
Completed | 242 | 266
Not Completed | 59 | 33
Not completed — Lost to Follow-up | 57 | 31
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention) | Total
Number analyzed (Participants) | 301 | 299 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11) | 64 (11) | 63 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 177 | 357
  Male | 121 | 122 | 243
Years since stroke [Mean (Standard Deviation); unit: years] | 1.8 (1.4) | 1.8 (1.5) | 1.8 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Percentage of Participants with Blood Pressure controlled at <140/90 mm Hg
Time Frame: 6 months post enrollment into trial
Measure: Number; unit: percentage of participants
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Number analyzed (Participants) | 242 | 266
percentage of participants | 76 | 65

2. Primary Outcome: LDL Cholesterol
Description: Percentage of participants with controlled Low Density Lipoprotein low (LDL) of less than 100 mg/dL
Time Frame: 6 months post enrollment into trial
Measure: Number; unit: percentage of participants
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Number analyzed (Participants) | 242 | 266
percentage of participants | 59 | 57

3. Primary Outcome: Use of Anti-thrombotic Medication
Description: Number of participants taking anti-thrombotic medication
Time Frame: 6 months post enrollment into trial
Measure: Number; unit: participants
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Number analyzed (Participants) | 242 | 266
participants | 199 | 226

4. Secondary Outcome: Knowledge and Attitudes About Stroke Recurrence Risk
Time Frame: 6 months post enrollment into trial
Reporting Status: Not Posted

5. Secondary Outcome: Medication Adherence
Description: Number of participants adherent to medications as determined with Morisky score ≥ 6 Adherence to medications was measured using the 8-item Morisky Medication Adherence Questionnaire (Morisky). The questionnaire has been validated against an objective measure of adherence and has been used in racially diverse and elderly patient samples. Scores on the questionnaire can be used to classify patients into low and high adherence groups.
  Consistent with standard cut points, participants who scored less than 6 points on the Morisky were categorized as nonadherent to medications and participants who scored 6 to 8 points were categorized as adherent.
Time Frame: 6 months post enrollment into trial
Measure: Number; unit: participants
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Number analyzed (Participants) | 242 | 266
participants | 159 | 169

6. Secondary Outcome: Emotional Health
Description: Number of participants diagnosed as depressed utilizing depression scale. Participant is determined to be depressed if Patient Health Questionnaire (PHQ8) ≥ 10. Scale has a total score between 0 and 24 points. A total score of 0 to 4 represents no significant depressive symptoms. A total score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe.
Time Frame: 6 months post enrollment into trial
Measure: Number; unit: participants
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Number analyzed (Participants) | 242 | 266
participants | 46 | 59

7. Secondary Outcome: Access to Medical Care
Description: Number of participants who have a primary care doctor
Time Frame: 6 months post enrollment into trial
Population: 1 missing response from Usual Care group
Measure: Number; unit: participants
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Number analyzed (Participants) | 242 | 265
participants | 232 | 240

ADVERSE EVENTS:
Arm/Group | Peer-Led Stroke Recurrence Prevention Education | Usual Care (Delayed Intervention)
Serious Adverse Events (participants affected / at risk) | 0/301 | 0/299
Other Adverse Events (participants affected / at risk) | 0/301 | 0/299

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes